CLINICAL TRIAL: NCT00450151
Title: Effect of Cardiopulmonary Bypass on Platelet Activation Markers Such as Platelet Factor 4 and Transforming Growth Factor B, in Pediatric Cardiac Surgery
Brief Title: Platelet Activation Markers in Pediatric Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Aarti Sharma, Associate Professor of Anesthesiology, Weill Medical College of Cornell University
Other Study IDs: 0612008895
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Coronary Disease
Keywords: Pediatric; Cardiopulmonary bypass Surgery; Cardiac Surgery; Platelet; Platelet Activation Markers; Platelet Factor4; Transforming Growth Factor Beta
MeSH Terms: conditions — Coronary Disease; Camurati-Engelmann Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For all patients, after obtaining written consent, 3.15ml of blood will be collected in CTAD tubes, from arterial line pre cardiopulmonary bypass and post cardiopulmonary bypass. Blood sample will be cooled in ice bath, centrifuged at 2500 rpm for 30 minutes, and supernatant plasma sample will be collected. This plasma will be stored at -20 degrees celcius or below. Enzyme-linked immunosorbent assay (ELISA) will be performed using the plasma to make quantitative assessment of platelet factor 4 and transforming growth factor beta.
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study the focus will be on correlating the levels of platelet activation markers (proteins that are released when blood cells are activated)to the duration of cardiopulmonary bypass, temperature during cardiopulmonary bypass and the weight of the patient.

DETAILED DESCRIPTION:
This research is being done because we would like to learn more about platelet dysfunction in children undergoing cardiopulmonary bypass.

It has been an established fact that cardiopulmonary bypass causes dysfunction in platelets. Activation of platelets during cardiopulmonary bypass is implicated as being a major factor in causing platelet dysfunction.

For all participants, approximately 3.15 ml of blood will be collected in special tubes called CTAD tubes, before and after cardiopulmonary bypass (6.30ml in total). This amount of blood draw is well within the guidelines of NIH (National Institute of Health).

Enzyme-linked immunosorbent assay (ELISA) will be performed using this plasma to make quantitative assessment of Platelet factor 4 and Transforming growth factor beta.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to have surgery involving cardiopulmonary bypass for congenital cardiac abnormalities.
* Age: Newborn to 7 years
* Gender: male and female

Exclusion Criteria:

* Emergency surgery
* Weight less than 3 kg
* Age greater than 7 years
* Patients with low platelet counts (<100,000)
* Patients on medications that are known to interfere with platelet function such as prostacyclins, non-steroidal anti-inflammatory drugs, plavix.

Patients whose parents not willing to give consent

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The targeted population will be pediatric patients with congenital heart defects who will be needing cardiopulmonary bypass (CPB) while undergoing cardiac surgery. The age range will be newborn to 7 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Sharma, MD, Principal Investigator — Weill Medical College-New York Presbyterian Hospital
Locations (1):
- NewYork-Presbyterian Hospital-Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Background] Garlichs CD, Eskafi S, Raaz D, Schmidt A, Ludwig J, Herrmann M, Klinghammer L, Daniel WG, Schmeisser A. Patients with acute coronary syndromes express enhanced CD40 ligand/CD154 on platelets. Heart. 2001 Dec;86(6):649-55. doi: 10.1136/heart.86.6.649. PMID 11711459
- [Background] Ichinose F, Uezono S, Muto R, Uchida H, Hatori F, Terui K, Niimi Y, Goto T, Nakata Y, Morita S. Platelet hyporeactivity in young infants during cardiopulmonary bypass. Anesth Analg. 1999 Feb;88(2):258-62. doi: 10.1097/00000539-199902000-00006. PMID 9972737
- [Background] Rinder CS, Bohnert J, Rinder HM, Mitchell J, Ault K, Hillman R. Platelet activation and aggregation during cardiopulmonary bypass. Anesthesiology. 1991 Sep;75(3):388-93. doi: 10.1097/00000542-199109000-00002. PMID 1716077